CLINICAL TRIAL: NCT01158079
Title: A Multi-center, Open-Label, Extension Study of ALN-VSP02 in Cancer Patients Who Have Responded to ALN-VSP02 Treatment
Brief Title: Multi-center, Open Label, Extension Study of ALN-VSP02 in Cancer Patients Who Have Responded to ALN-VSP02 Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-VSP02-002
Record Dates: First submitted 2009-12-11; First posted 2010-07-08 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Solid Tumors
Keywords: Liver; Solid Tumors; Advanced Solid Tumors with Liver Involvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ALN-VSP02 — The dose of ALN-VSP02 will be administered at the same dose level and schedule received at the completion of the previous study

SUMMARY:
This study provides a mechanism for continued administration of ALN-VSP02 therapy to patients with cancer who completed participation in another ALN-VSP02 clinical study. The primary objective of this study is to collect long term safety data.

DETAILED DESCRIPTION:
Study ALN-VSP02 is an extension study for previously conducted ALN-VSP02 studies. The study is being conducted to allow for continued ALN-VSP02 therapy for patients who completed participation in an ALN-VSP02 clinical study, achieved clinical benefit with ALN-VSP02 (i.e., disease response of stable disease or better), and, in the Investigator's opinion, may benefit from continuation of ALN-VSP02 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has completed a previous ALN-VSP02 study, and is deemed to have stable disease or better.
2. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
3. Patient has adequate hematologic, liver, and renal function.

Exclusion Criteria:

1. Patient is receiving full-dose (therapeutic) anticoagulation therapy and/or aspirin > 325 mg/day or other platelet inhibitory agents.
2. Patient has clinically significant cardiovascular disease or uncontrolled serious cardiac arrhythmia.
3. Patient has clinically significant cerebrovascular disease.
4. Patient has a seizure disorder not controlled on medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Collect long term ALN-VSP02 safety data | Throughout the study
  Patients remain on treatment until disease progression or an adverse event. Adverse events are assessed throughout treatment.

SECONDARY OUTCOMES:
Assess disease response by Response Evaluation Criteria In Solid Tumors (RECIST) | Every 2 months
  Disease response is assessed every 2 months until the patient stops treatment due to disease progression or an adverse event
Evaluate preliminary evidence of antitumor activity/antiangiogenic activity | Every 3 - 6 months
  Evaluations will take place every 3-6 months until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Vaishnaw, MD PhD, Study Director — Alnylam Pharmaceuticals
Locations (10):
- United States (7):
  - TGen Clinical Research Service at Scottsdale Healthcare, Scottsdale, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Spain (3):
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia